CLINICAL TRIAL: NCT02061241
Title: Intracardiac Haemo-dynamics and Echocardiographic Assessment to Optimise Lead Placement for CRT
Brief Title: A Comparison of Two Techniques for Choosing the Best Place to Put a Pacing Lead for Cardiac Resynchronisation Therapy
Acronym: IDEAL-CRT
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Dr James Gamble, Co-investigator, Oxford University Hospitals NHS Trust
Other Study IDs: NIHR CSP 146533; 14/SC/0148 (Other: UK NRES)
Record Dates: First submitted 2014-02-07; First posted 2014-02-12 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
Keywords: Cardiac resynchronisation therapy; Pacing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients: All included patients, having CRT implant procedure Will have both Pacing in vein at site of latest mechanical activation and Pacing in other suitable vein.
  Interventions: Procedure: Pacing in vein at site of latest mechanical activation; Procedure: Pacing in other suitable vein

INTERVENTIONS:
Procedure: Pacing in vein at site of latest mechanical activation — Pacing in vein at site of latest mechanical activation
Procedure: Pacing in other suitable vein — Pacing in other suitable vein

SUMMARY:
Cardiac resynchronisation therapy (CRT) using biventricular pacing (BiVP) is established as an effective treatment for heart failure. Unfortunately up to 45% of patients do not respond, with no improvement in symptoms or cardiac size. Reducing the proportion of non-responders has become the key research focus in CRT.

Targeting the position of the left ventricular (LV) pacing lead within the coronary vein network has previously been shown to increase the proportion of responders to CRT. Several techniques have been tried for targeting lead position, of which the best investigated are the use of speckle-tracking echocardiography to target the lead position to the site of latest mechanical activation of the left ventricle, and the use of invasive monitoring to select the pacing site at which the greatest acute haemodynamic response (AHR) to BiVP occurs. Both techniques are limited by groups of patients in whom the techniques are not possible or provide limited useful information.

The relationship between these two measures is unknown - there are no previous studies that have investigated correlation between the site of latest mechanical activation determined by echo and the site of maximal AHR. It is likely that a hybrid technique using both of these investigations might allow optimal lead positioning in more patients, or that if the information is shown to be equivalent, more streamlined techniques can be designed.

This study will also be able to contribute towards several important secondary questions. In particular the investigators will study the possibility of using non-invasive cardiac output monitoring (NICOM) to assess haemodynamic response rather than an intravascular pressure monitor wire. The investigators also wish to assess whether the site of latest mechanical activation is changed by right ventricular pacing.

ELIGIBILITY:
Inclusion Criteria:

* With ejection fraction <35%
* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Indication for cardiac resynchronisation therapy

Exclusion Criteria:

* Left Ventricular Ejection Fraction >35%
* Severe peripheral vascular disease (that would make arterial access more risky)
* Haemodynamic instability (such that a longer procedure is inadvisable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Due to have CRT device implants.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Acute haemodynamic response in area of latest mechanical activation and another vein | Time 0 (during implant procedure)
  To assess whether pacing at the site of latest mechanical activation produces the maximal acute haemodynamic response to biventricular pacing, when compared to other attainable Left Ventricular coronary venous pacing sites.
  Acute haemodynamic response measured as percentage change in left ventricular dP/dt max (maximum rate of change of left ventricular pressure) recorded by a left ventricular pressure wire, between baseline atrial pacing at 80 beats per minute and biventricular pacing in each vein

SECONDARY OUTCOMES:
Maximum acute haemodynamic response between all available pacing vectors in the vein within the area of latest mechanical response | Time 0 (during implant procedure)
  To assess if further increases in acute haemodynamic response at the site of latest mechanical activation can be achieved with different pacing configurations.
Acute haemodynamic response by NICOM and pressure wire | Time 0 (during implant procedure)
  To compare results attained from non-invasive cardiac output monitoring (NICOM) to those from invasive monitoring
Area of latest mechanical activation in right ventricular pacing and intrinsic rhythm | 1 day post procedure
  To assess the effect of right ventricular pacing on the site of latest mechanical activation. Assessed using speckle-tracking echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Tim R Betts, MBChB, MD, Principal Investigator — Oxford University Hospitals
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Khan FZ, Virdee MS, Palmer CR, Pugh PJ, O'Halloran D, Elsik M, Read PA, Begley D, Fynn SP, Dutka DP. Targeted left ventricular lead placement to guide cardiac resynchronization therapy: the TARGET study: a randomized, controlled trial. J Am Coll Cardiol. 2012 Apr 24;59(17):1509-18. doi: 10.1016/j.jacc.2011.12.030. Epub 2012 Mar 7. PMID 22405632
- [Background] McAlister FA, Ezekowitz J, Hooton N, Vandermeer B, Spooner C, Dryden DM, Page RL, Hlatky MA, Rowe BH. Cardiac resynchronization therapy for patients with left ventricular systolic dysfunction: a systematic review. JAMA. 2007 Jun 13;297(22):2502-14. doi: 10.1001/jama.297.22.2502. PMID 17565085
- [Background] Saba S, Marek J, Schwartzman D, Jain S, Adelstein E, White P, Oyenuga OA, Onishi T, Soman P, Gorcsan J 3rd. Echocardiography-guided left ventricular lead placement for cardiac resynchronization therapy: results of the Speckle Tracking Assisted Resynchronization Therapy for Electrode Region trial. Circ Heart Fail. 2013 May;6(3):427-34. doi: 10.1161/CIRCHEARTFAILURE.112.000078. Epub 2013 Mar 8. PMID 23476053
- [Background] Duckett SG, Ginks M, Shetty AK, Bostock J, Gill JS, Hamid S, Kapetanakis S, Cunliffe E, Razavi R, Carr-White G, Rinaldi CA. Invasive acute hemodynamic response to guide left ventricular lead implantation predicts chronic remodeling in patients undergoing cardiac resynchronization therapy. J Am Coll Cardiol. 2011 Sep 6;58(11):1128-36. doi: 10.1016/j.jacc.2011.04.042. PMID 21884950